CLINICAL TRIAL: NCT00002011
Title: The Therakos UVAR Photopheresis System in the Treatment of AIDS-Related Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Therakos (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 049A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-07

CONDITIONS: HIV Infections
Keywords: PUVA Therapy; Methoxsalen; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Methoxsalen

INTERVENTIONS:
Drug: Methoxsalen

SUMMARY:
To determine the safety and patient tolerance of UVAR Photopheresis System (extracorporeal photopheresis) in the Treatment of AIDS-Related Complex (ARC).

DETAILED DESCRIPTION:
Treatment involves the patient ingesting 8-methoxsalen (8-MOP) by mouth approximately two hours prior to each photopheresis session. The photopheresis instrument will separate the patient's white blood cells and some plasma from other blood components and return the majority of blood components to the patient. The separated white blood cells and plasma will be exposed to UVA (Ultraviolet A) light while outside the body. The UVA light photoactivates the 8-MOP drug which is now located in the DNA of the collected cells. After this exposure, the patients photoactivated white blood cells will be returned to the patient by venous access.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Diagnosis of AIDS-related complex (ARC).
* Veins that can provide adequate access.
* Negative drug screen for drugs of abuse and zidovudine (AZT).
* Be willing to adhere to the protocol and sign a patient informed consent prior to study entry.
* Live within adequate commuting distance to the treatment center.
* Not be on any other investigational drug/device.
* Be 18 - 80 years old but minimum age requirements may be affected by state regulations or specific medical conditions.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Inability to tolerate extracorporeal volume loss during the leukocyte-enrichment phase.
* Photosensitive disease, such as porphyria or systemic lupus erythematosus. Care must be taken in selecting patients who require drugs (either systemically or topically) during the course of the study with photosensitizing potential such as phenothiazines, tetracyclines, sulfonamides or chlorothiazide.
* Renal insufficiency with creatinine > 3 mg/dl.
* Symptoms of toxic effects (World Health Organization Criteria) resulting from previous therapy.
* Severe emotional, behavioral or psychiatric problems that in the opinion of the investigator would result in poor compliance with the treatment regimen.
* Idiosyncratic or hypersensitivity reactions to 8-MOP compounds.
* History of or active Pneumocystis carinii pneumonia, other opportunistic infection or neoplasms (Kaposi's sarcoma), or wasting syndrome.
* Active hepatitis.
* Aphakia because of the significantly increased risk of retinal damage due to absence of lenses.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Photosensitizing drugs should not be administered prior to photopheresis treatment.
* Other investigational drugs.

Concurrent Treatment:

Excluded:

* Other treatment using an investigational device.

Patients with the following are excluded:

* Inability to tolerate extracorporeal volume loss during the leukocyte-enrichment phase.
* Photosensitive disease.
* Symptoms of toxic effects (World Health Organization Criteria) resulting from previous therapy.
* Severe emotional, behavioral or psychiatric problems that in the opinion of the investigator would result in poor compliance with the treatment regimen.
* Idiosyncratic or hypersensitivity reactions to 8-MOP compounds.
* Actively involved in drug abuse.
* Aphakia because of the significantly increased risk of retinal damage due to absence of lenses.

Prior Medication:

Excluded:

* Zidovudine (AZT).

Actively involved in drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Memorial Hosp, Morristown, New Jersey, United States